CLINICAL TRIAL: NCT01335568
Title: Intracorporeal Autologous Hepatocyte Matrix Implant: A New Tissue Engineering Procedure for Treatment of Hepatic Disease
Brief Title: Hepatocyte Matrix Implant Study Indonesia
Acronym: HMIIndo
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baermed (Other)
Responsible Party: Hans U. Baer, RS Gading Pluit, Universitas Tarumanagara Indonesia and Baermed Switzerland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Baermed 002
Record Dates: First submitted 2011-04-11; First posted 2011-04-14 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Liver Cirrhosis; Liver Insufficiency; Chronic Liver Disease
Keywords: Hepatocyte; Scaffold; Matrix; Liver cirrhosis; Liver insufficiency
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgery (Experimental): chronic liver insufficiency, cirrhosis
  Interventions: Procedure: Hepatocyte Matrix Implant

INTERVENTIONS:
Procedure: Hepatocyte Matrix Implant — Open surgical procedure with biopsy of liver tissue and pancreatic tissue for proceeding in institutional GMP laboratory. Implantation of autologous hepatocytes and islet cells on scaffolds into the small bowel mesentery. Usually 10 to 20 implants are used.
  Other Names: Hepatocyte matrix implantation; Hepatocyte scaffold implantation; Cell matrix implant

SUMMARY:
This clinical investigation of the hepatocyte matrix implant is an evaluation blinded non-randomized and monocentric pilot study of Phase I, which is conducted as a therapeutic investigation. Randomization is not possible due to ethical and practical reasons. This study has already been approved in Switzerland and has been adapted to Indonesian Law and disease.

This new treatment procedure has already been successfully used on the basis of compassionate use in Germany. The hepatocyte matrix implant is a new patented procedure consisting of bio-matrix technology. A formaldehyde-free special matrix consisting of self-dissolving polymers is applied as a carrier substance and is cultivated with human autologous cells using a special technique. Clinically the bio artificial liver replacement tissue for patients with end-stage hepatic disease has been developed as a first application. In this procedure autologous hepatocytic tissue and pancreatic tissue is removed (liver resection and pancreatic biopsy) from the patient in a first surgical procedure. The tissue is sent to a specialized Cell Culture Laboratory. The laboratory is GMP certified for this procedure. The cells are processed according to SOPs in a special perfusion procedure and prepared on several platelets of matrices (platelets of 20 mm diameter and 4mm thickness). After completion of the laboratory process the bio tissues are implanted into the mesentery of the small intestine during a second operation. The cells are growing controlled on the matrix, take on the capillaries of the patient and thus connect to the blood circulation. The implanted cells multiply by a specific factor and independently take over the metabolic function of the original liver after two to four weeks. In the following process the carrier matrix dissolves completely and implanted cells develop into liver cell tissue.

DETAILED DESCRIPTION:
This new treatment procedure has already been successfully used on the basis of individual treatment in Germany. The hepatocyte matrix implant is a new patented procedure consisting of bio-matrix technology. A formaldehyde-free special matrix consisting of self-dissolving polymers is applied as a carrier substance and is cultivated with human autologous cells using a special technique. Clinically the bio artificial liver replacement tissue for patients with end-stage hepatic disease has been developed as a first application. In this procedure autologous hepatocytic tissue and pancreatic tissue is removed (liver resection and pancreatic biopsy) from the patient in a first surgical procedure. The tissue is sent to a specialized Cell Culture Laboratory. The laboratory is GMP certified for this procedure. The cells are processed according to SOPs in a special perfusion procedure and prepared on several platelets of matrices (platelets of 20 mm diameter and 4mm thickness). After completion of the laboratory process the bio tissues are implanted into the mesentery of the small intestine during a second operation. The cells are growing controlled on the matrix, take on the capillaries of the patient and thus connect to the blood circulation. The implanted cells multiply by a specific factor and independently take over the metabolic function of the original liver after two to four weeks. In the following process the carrier matrix dissolves completely and implanted cells develop into liver cell tissue.

ELIGIBILITY:
Inclusion Criteria:

* endstage liver disease
* stable and non-improving liver condition for at least 3 month
* alcoholic liver cirrhosis: proven alcohol abstinence for 6 month or more
* patient in bad general condition

Exclusion Criteria:

* pregnancy
* drug addiction (except alcohol)
* psychiatric disease
* HIV positive
* sepsis
* peritoneal carcinosis
* hereditary liver disease
* acute liver failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical and laboratory parameters of liver function | 6 months
  Evaluation of clinical parameters MELD, CHILD, Asictes, portal hypertension in comparison of values measured 3 and 6 months before operation Evaluation of laboratory parameters Bilirubin, ASAT, ALAT, alkaline phosphatase, cholinesterase, albumin, total protein

CONTACTS AND LOCATIONS:
Overall Officials: Hans U Baer, Prof, MD, Principal Investigator — Baermed, RS Gading Pluit, UNTAR
Locations (1):
- R.S. Gading Pluit, Jakarta, Indonesia

REFERENCES:
- [Derived] Hendrawan S, Lheman J, Nuraeni, Weber U, Baer HU. Hepatocyte and Islet Cell Cotransplantation on Poly-L-Lactide Matrix for the Treatment of Liver Cirrhosis. Int J Hepatol. 2020 Oct 13;2020:5410359. doi: 10.1155/2020/5410359. eCollection 2020. PMID 33123384
- See also: Baermed Centre for Abdominal Surgery, Zurich, Switzerland — http://baermed.ch